CLINICAL TRIAL: NCT05023382
Title: Special Drug Use Investigation of Revestive Subcutaneous Injection 3.8 mg (All-case Surveillance)
Brief Title: A Study of Teduglutide in Japanese People With Short Bowel Syndrome
Status: Recruiting | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: TAK-633-5001; jRCT2031210284 (Registry Identifier: jRCT)
Record Dates: First submitted 2021-08-23; First posted 2021-08-26 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Short Bowel Syndrome
MeSH Terms: conditions — Short Bowel Syndrome | interventions — teduglutide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Teduglutide 0.05 milligram per kilogram (mg/kg): Participants will receive Teduglutide 0.05 milligram per kilogram (mg/kg) subcutaneous (SC) injection once daily.
  Interventions: Drug: Teduglutide

INTERVENTIONS:
Drug: Teduglutide — Teduglutide 0.05 mg/kg SC injection
  Other Names: TAK-633; Revestive

SUMMARY:
The main aims of this study are to check for side effects from treatment with teduglutide (Revestive) and how well teduglutide controls symptoms of short bowel syndrome.

The study sponsor will not be involved in how the participants are treated but will provide instructions on how the clinics will record what happens during the study.

During the study, participants with short bowel syndrome will receive an injection of teduglutide just under the skin (subcutaneous) according to their clinic's standard practice. The study doctors will check for side effects from teduglutide for 36 months.

ELIGIBILITY:
Inclusion Criteria:

* All participants in Japan who received teduglutide will be enrolled in this post marketing surveillance.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All participants in Japan who received teduglutide will be enrolled in this post marketing surveillance.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events | Up to 36 months
  An adverse event (AE) is any untoward or undesirable medical occurrence in a participant linked in time with the use of a pharmaceutical/ medicinal product. They are not limited to the events with clear causal relationship with treatment with concerned drug. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not related to the medicinal product.
Number of Participants with Serious Adverse Events | Up to 36 months
  A serious AE is any untoward medical occurrence or effect that at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability /incapacity, is a congenital anomaly / birth defect or is medically important due to other reasons than the above mentioned criteria.

SECONDARY OUTCOMES:
Changes from Baseline in Prescription Volume of Parenteral Nutrition Intravenous (PN/IV) Support | Baseline, 6, 12, 18, 24, 30, and 36 months after teduglutide treatment initiation
  Changes from baseline in prescription volume of PN/IV support prescribed by investigators to 6, 12, 18, 24, 30, and 36 months after teduglutide treatment initiation will be reported.
Percent Change from Baseline in Prescription Volume of PN/IV Support | Baseline, 6, 12, 18, 24, 30, and 36 months after teduglutide treatment initiation
  Percent change from baseline in prescription volume of PN/IV support to multiple timepoints (6, 12, 18, 24, 30, and 36 months) after teduglutide treatment initiation will be reported. Percent change from baseline will be calculated as following; [prescription volume at each timepoint - prescription volume at baseline] / prescription volume at baseline * 100 (percent).
Changes from Baseline in Dose of PN/IV Support | Baseline, 6, 12, 18, 24, 30, and 36 months after teduglutide treatment initiation
  Changes from baseline in actual dose of PN/IV support to 6, 12, 18, 24, 30, and 36 months after teduglutide treatment initiation will be reported.
Percent Change from Baseline of Dose in PN/IV Support | Baseline, 6, 12, 18, 24, 30, and 36 months after teduglutide treatment initiation
  Percent change from baseline in actual dose of PN/IV support to multiple timepoints (6, 12, 18, 24, 30, and 36 months) after teduglutide treatment initiation will be reported. Percent change from baseline will be calculated as following; [actual dose at each timepoint - actual dose at baseline] / actual dose at baseline * 100 (percent).
Percentage of Participants who Completely Wean off PN/IV Support | Baseline, 6, 12, 18, 24, 30, and 36 months after teduglutide treatment initiation
  Number of participants who completely wean off PN/IV support will be assessed.
Crohn's Disease Activity Index (CDAI) | 36 months after teduglutide treatment initiation
  CDAI score is calculated from the following 8 items: (a) Number of liquid or very soft stools; (b) Abdominal pain; (c) General wellbeing; (d) Extraintestinal complications; (e) Antidiarrhoeal drugs; (f) Abdominal mass; (g) Hematocrit; and (h) Body weight. Scores of some items in CDAI are calculated based on patient diary. Total range of score is more than 0. Higher score means more severe disease and especially severe disease was defined as a value of greater than 450.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (2):
- Japan (2):
  - Takeda Selected Site, Tokyo, Tokyo
  - Takeda selected site, Tokyo, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Wada M, Nakamura S, Hayashi A, Otake R, Miyamoto M, Tanaka T. Six-Month Safety and Effectiveness of Teduglutide in Patients with Short Bowel Syndrome in Japan: Interim Analysis of Post-marketing Surveillance. Adv Ther. 2026 Jan;43(1):425-441. doi: 10.1007/s12325-025-03398-y. Epub 2025 Dec 1. PMID 41324792
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/612d4d9dc61629002b6311cb